CLINICAL TRIAL: NCT05086445
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3502970 in Japanese Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3502970 in Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17610; J2A-JE-GZGB (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-20; First posted 2021-10-21 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3502970 (Part A) (Experimental): Single doses of LY3502970 administered orally.
  Interventions: Drug: LY3502970
- LY3502970 (Part B) (Experimental): Multiple doses of LY3502970 administered orally.
  Interventions: Drug: LY3502970
- Placebo (Part A) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3502970 — Administered orally
  Arms: LY3502970 (Part A); LY3502970 (Part B)
Drug: Placebo — Administered orally
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to learn about the side effects of LY3502970 when given to Japanese participants with type 2 diabetes mellitus (T2DM). Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. For each participant, the study will last up to 24 weeks, inclusive of screening and will include 10 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Males and females not of childbearing potential
* Have type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year
* Have glycated hemoglobin (HbA1c) value ≥ 7.0% and ≤ 10.0% for participants treated with diet and exercise or HbA1c ≥ 6.5% and ≤ 9.0% for participants who have washed out antidiabetic medications at screening
* Have type 2 diabetes controlled with diet and exercise alone or are stable on a single oral antidiabetic medication (OAM); either metformin, DPP-4 (dipeptidyl peptidase-4) inhibitor, or SGLT2 (sodium-glucose co-transporter-2) inhibitor within 3 months prior to screening. Participants must withdraw from their OAM treatment for at least 28 days prior to dosing.

Exclusion Criteria:

* Have type 1 diabetes mellitus or latent autoimmune diabetes in adults.
* Have uncontrolled diabetes defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization
* Have had an episode of severe hypoglycemia, as defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery or have a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms.
* Have a history of acute or chronic pancreatitis or fasting serum triglyceride level of >500 milligram per deciliter (mg/dL).
* Have known liver disease, obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aminotransferases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 3× upper limit of normal (ULN).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 15
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3502970 | Predose on Day 1 through up to Day 88
  PK: Cmax of LY3502970
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3502970 | Predose on Day 1 through up to Day 88
  PK: AUC of LY3502970
Change from Baseline in Fasting Glucose | Baseline through Day 85
  Change from Baseline in Fasting Glucose
Change from Baseline in Glycated Hemoglobin (HbA1c) | Baseline through Day 85
  Change from Baseline in HbA1c
Change from Baseline in Body Weight | Baseline through Day 88
  Change from Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Japan (5):
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - P-One Clinic, Hachiōji, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Medical Corporation Houeikai Sekino Clinical Pharmacology Clinic, Toshima City, Tokyo
  - Yokohama Minoru Clinic, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3502970 in Japanese Participants With Type 2 Diabetes Mellitus — https://trials.lillytrialguide.com/en-US/trial/19e2wyNokvTUEXgJp8UDry